CLINICAL TRIAL: NCT06712225
Title: Combining Anomia Therapy and Executive Function Training in Chronic Post-stroke Aphasia: a Pilot Study of Multidimensional Effects
Brief Title: Anomia Therapy and Executive Function Training in Chronic Post-stroke Aphasia: Pilot Study of Multidimensional Effects
Acronym: ATAC2PILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL22_0566
Record Dates: First submitted 2024-10-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Aphasia, Acquired; Speech Therapy
Keywords: Post-stroke aphasia; Speech-therapy; Anomia therapy; Executive function; Discourse; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Aphasia; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Anomia Therapy alone (Active Comparator)
  Interventions: Behavioral: Anomia therapy: semantic feature analysis and phonological components analysis;
- Arm B: Anomia Therapy + Executive Function Training (Experimental)
  Interventions: Behavioral: Anomia therapy: semantic feature analysis and phonological components analysis;; Behavioral: Executive function training: computerized equipment

INTERVENTIONS:
Behavioral: Anomia therapy: semantic feature analysis and phonological components analysis; — After the initial assessment + functional Magnetic Resonance Imaging (fMRI), participants will first receive their usual speech therapy rehabilitation for 10 to 15 sessions (baseline phase), and then enter the experimental phase: 18 sessions (3 per week) of either anomia therapy alone or anomia therapy + executive function training, according to the arm they were assigned to. All sessions will last 45 minutes. Naming skills will be repeatedly measured during both phases. A second assessment of language + fMRI will then be conducted and participants will return to their usual rehabilitation. Four weeks later, a final assessment of naming and discourse will be conducted.
Behavioral: Executive function training: computerized equipment — Executive function training will be conducted by means of a computerized material specifically designed for the study, consisting of verbal and nonverbal exercises targeting, always in the same order, inhibition, shifting, working memory and planning functions, with a gradient of difficulty. Training will always be done at the beginning of the session, during 20 minutes, before anomia therapy.
  Arms: Arm B: Anomia Therapy + Executive Function Training

SUMMARY:
The goal of this clinical trial is to measure the effects of a speech therapy protocol combining anomia therapy and executive function training on naming and discourse in people with chronic aphasia, and to study the related brain changes.

The main questions it aims to answer are:

* Does the protocol improve naming skills ?
* Do the improvements observed transfer to discourse abilities ?
* Are there any brain changes induced by this protocol ?

Researchers will compare anomia therapy alone to anomia therapy + executive function training to see if the latter works better.

Participants will:

* Have a whole language assessment and a Magnetic Resonance Imaging (MRI) scan in the hospital before and after the protocol
* Receive 18 sessions of the protocol, 3 times a week during 6 weeks, in the hospital
* Have several naming assessments during the protocol

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-80 years old) with post-stroke aphasia (> 6 months post-stroke)
* Participant or legal representative able to understand the aims of the study
* Participant or legal representative who have signed an informed consent form

Exclusion Criteria:

* Aphasia with severe anarthria (mutism), comprehension disorders or alexia, incompatible with the purpose of the study
* Contraindications for MRI
* History of head trauma, brain tumor, neurodegenerative disease, or any other neurological or psychiatric condition
* Non-affiliation to social welfare

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in repeated measures of naming scores | Every 2 or 3 sessions during the baseline phase (3 sessions per week during 3,5 to 5 weeks) and during the experimental phase (3 sessions per week during 6 weeks)
  Naming skills will be repeatedly assessed for each participant every 2 or 3 sessions during the 3,5 to 5 weeks of the baseline phase (usual rehabilitation): 5 to 7 measures, and during the 6 weeks of the experimental phase: 6 to 9 measures. A naming task specifically designed for the study ("Deno 100"), including 100 black and white line drawing pictures will be used to this end. Scores will range from 0 (no item correctly named) to 100 (all items correctly named). A visual analysis (mean and trend) and statistical analyses will then be applied in order to measure the effect of the experimental treatment on treated words and the effect size.

SECONDARY OUTCOMES:
Comparison of pre and post intervention control naming scores for each group (arm A / arm B) and between groups. | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, 6 weeks after: just after the intervention, and 4 weeks after
  In order to measure the effects of the experimental treatment on non-treated words (transfer), a control naming task (French Battery of lexical disorders assessment, score range [0-54]) will be administered to each participant. Mean scores will be compared for each group at several times, and between groups at each time.
Comparison of pre and post intervention discourse scores for each group (arm A / arm B) and between groups: Productivity (number of words produced / minute) | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, and 4 weeks after the intervention
  In order to measure the effects of the experimental treatment on discourse abilities (transfer), five samples of discourse will be collected from each participant (two picture descriptions, one wordless picture book-supported narrative, one personal narrative and one procedural information). Different scores will be calculated: productivity (number of words produced / min), informativity (% of correct information units), lexical diversity (type-token ratio), syntactic structure (Predicate Argument Structure), and efficience (Main Concept Analysis). These scores will be compared for each group at several times, and between groups at each time.
Comparison of pre and post intervention discourse scores for each group (arm A / arm B) and between groups: Informativity (% of correct information units) | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, and 4 weeks after the intervention
  In order to measure the effects of the experimental treatment on discourse abilities (transfer), five samples of discourse will be collected from each participant (two picture descriptions, one wordless picture book-supported narrative, one personal narrative and one procedural information). Different scores will be calculated: productivity (number of words produced / min), informativity (% of correct information units), lexical diversity (type-token ratio), syntactic structure (Predicate Argument Structure), and efficience (Main Concept Analysis). These scores will be compared for each group at several times, and between groups at each time.
Comparison of pre and post intervention discourse scores for each group (arm A / arm B) and between groups: Lexical diversity (type-token ratio) | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, and 4 weeks after the intervention
  In order to measure the effects of the experimental treatment on discourse abilities (transfer), five samples of discourse will be collected from each participant (two picture descriptions, one wordless picture book-supported narrative, one personal narrative and one procedural information). Different scores will be calculated: productivity (number of words produced / min), informativity (% of correct information units), lexical diversity (type-token ratio), syntactic structure (Predicate Argument Structure), and efficience (Main Concept Analysis). These scores will be compared for each group at several times, and between groups at each time.
Comparison of pre and post intervention discourse scores for each group (arm A / arm B) and between groups: Syntactic structure (Predicate Argument Structure) | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, and 4 weeks after the intervention
  In order to measure the effects of the experimental treatment on discourse abilities (transfer), five samples of discourse will be collected from each participant (two picture descriptions, one wordless picture book-supported narrative, one personal narrative and one procedural information). Different scores will be calculated: productivity (number of words produced / min), informativity (% of correct information units), lexical diversity (type-token ratio), syntactic structure (Predicate Argument Structure), and efficience (Main Concept Analysis). These scores will be compared for each group at several times, and between groups at each time.
Comparison of pre and post intervention discourse scores for each group (arm A / arm B) and between groups: Efficience (Main Concept Analysis) | First day of the baseline phase, 3,5 to 5 weeks after: first day of the experimental phase, and 4 weeks after the intervention
  In order to measure the effects of the experimental treatment on discourse abilities (transfer), five samples of discourse will be collected from each participant (two picture descriptions, one wordless picture book-supported narrative, one personal narrative and one procedural information). Different scores will be calculated: productivity (number of words produced / min), informativity (% of correct information units), lexical diversity (type-token ratio), syntactic structure (Predicate Argument Structure), and efficience (Main Concept Analysis). These scores will be compared for each group at several times, and between groups at each time.
MRI: Quantitative analyses | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  Location of the cerebral vascular accident (3DT1) and analysis of lesion volumes (3D FLAIR)
MRI: Qualitative analyses | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  Functional connectivity:
  Task-based functional MRI (Naming, phonological and semantic processes); Rest-based functional MRI

OTHER OUTCOMES:
Aphasia profile and severity score | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  The aphasia profile and severity score will be determined by means of the Quick Aphasia Battery. Scores range from 0 to 10: < 5 = severe aphasia; 5 to 7,5 = moderate aphasia; 7,5 to 8,9 = mild aphasia
Semantic association | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  Semantic processing will be assessed by means of the semantic association task of the French Battery of lexical disorders assessment, in which the participant is asked to match semantically related pictures (score range [0-54])
Executive function: Modified Card Sorting Test | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  The Modified Card Sorting Test explores flexibility, inhibition, updating and attention skills through a card sorting task following 3 rules: colour, number and shape.
Executive function: Verbal fluency | Before the baseline and just after the intervention: 9,5 to 11 weeks after
  Each participant will be asked to produce words beginning with the letter /p/ in 2 minutes and then names of animals during 2 minutes. The number of words produced in each category will be compared with French norms (Grefex)
Questionnaire of Quality of Life | Before the baseline and 4 weeks after the intervention
  In order to measure the functional effects of the experimental treatment, a quality of life scale (Stroke and Aphasia Quality of Life scale: score ranging from 1: low quality of life to 39: good quality of life) will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MORITZ-GASSER, Pr, Principal Investigator — University Hospital, Montpellier